CLINICAL TRIAL: NCT05711888
Title: A Sensitive Measurement Proposal in Alzheimer's Disease: Semantic Recognition Task
Brief Title: Semantic Recognition Task (SRT) in Alzheimer Disease
Acronym: SRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Jbid DURSUN UNCU, PhD Student, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-29624016-050.99-1484553
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Recognition; Semantic; Memory; Free and Cued Selective Reminding Test
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Semantic recognition task outcomes are observed in people diagnosed with Alzheimer's disease with Non-Alzheimer population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Semantic information in Alzheimer Disease (Experimental): To observe the semantic information processing in early stages of Alzheimer Disease is the main aim of the study. A paper-pencil neuropsychological assessment battery will be used. For memory testing FCSRT (free and cued selective reminding test) will be used. The patients are going to be assessed while in clinical diagnosis routine.
  Interventions: Behavioral: Semantic Recognition Procedure

INTERVENTIONS:
Behavioral: Semantic Recognition Procedure — A semantic recognition task is going to be added to administrated FCSRT procedure after immediate and delayed recall phases.

SUMMARY:
The goal of this study is to observe the outcomes of a semantic recognition task in Alzheimer Disease and discuss what this might add to clinical practice.

DETAILED DESCRIPTION:
In classical memory testing procedures, the outcomes of recognition task is related to hippocampal memory deficits knowing that the recognition task is not purely temporal lobe activity. The aim of this study is to propose a recognition task more specific to temporal lobe activity.

ELIGIBILITY:
Inclusion Criteria:

* to have biomarker analysis for Alzheimer disease (positive or negative).

Exclusion Criteria:

* illiteracy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2027-12-26 (Estimated)

PRIMARY OUTCOMES:
Semantic Recognition Task | 1 day
  The number of correct answers will be observed just after the short-term learning procedure and just after the delayed recall procedure among people with positive biomarker compared to those with negative biomarker to Alzheimer Disease.

CONTACTS AND LOCATIONS:
Overall Officials: İ. Hakan Gürvit, Prof. MD., Study Director — Istanbul University
Locations (1):
- Jbid Dursun Uncu, Beşiktaş, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No